CLINICAL TRIAL: NCT03615508
Title: Exploration of Pupil Dilation in Horner's Patients Taking Flomax
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: incomplete enrollment
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Cristos Ifantides, MD, MBA, Associate Professor, Department of Ophthalmology, Denver Health and Hospital Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COMIRB 18-0620
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Horner Syndrome
Keywords: Alpha blockers; Tamsulosin
MeSH Terms: conditions — Horner Syndrome | interventions — Phenylephrine

STUDY DESIGN:
Intervention Model Description: Single arm, intervention trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 10% phenylephrine (Other): All patients will receive 10% phenylephrine at their eye examination as the drug to dilate the pupil. After pupil dilation, pupil size will be measured.
  Interventions: Drug: 10% phenylephrine

INTERVENTIONS:
Drug: 10% phenylephrine — 10% phenylephrine is a drug that can be used to dilate patient's eyes at their yearly eye examination. All enrolled subjects will receive this drug for their eye dilation.
  Other Names: Phenylephrine 10%, Pupil Dilation

SUMMARY:
This study is evaluating the pupil dilation of Horner's Patients who have ever taken an alpha blocker such as Tamsulosin. Patients will undergo eye dilation as would occur at a yearly eye examination, but their pupil dilation measurements will be recorded.

DETAILED DESCRIPTION:
This study will enroll 10 participants who have a unilateral Horner's Syndrome AND have a history of taking an alpha blocker such as Tamsulosin. Participants will be recruited based on those two enrollment criteria, and after consenting they will undergo pupil dilation with 10% phenylephrine. Once fully dilated the pupil size will be measured. Pupil dilation size of the eye affected by the Horner's Syndrome will be compared to the eye not affected by Horner's. Primary study outcome is the comparative dilation size of the Horner's affected eye to the non affected eye in all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Horner's Syndrome
2. History of taking an alpha blocker (tamsulosin/ terazosin/doxazosin/alfuzosin/silodosin) medication

Exclusion Criteria:

1. Subjects with untreated hypertension
2. Subjects with thyrotoxicosis
3. Pregnant women
4. Prisoners
5. Inability to consent
6. Subjects with anatomical narrow angles who have never had a dilated exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristos Ifantides, MD, Principal Investigator — Denver Health
Locations (2):
- United States (2):
  - University of Colorado Hospital, Rocky Mountain Lions Eye Institute, Denver, Colorado
  - Denver Health, Denver, Colorado

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 10% Phenylephrine
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study terminated, no patients analyzed; Data not reported for 1 participant for privacy reasons.
Arm/Group | 10% Phenylephrine
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Pupil Size Measurements
Description: pupil dilation measurements will be taken of each eye at the eye examination.
Time Frame: 20-30 minutes after 10% phenylephrine has been placed in each eye.
Population: Study incomplete. Only 1 subject enrolled and data not reported for 1 participant for privacy reasons.
Arm/Group | 10% Phenylephrine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: N/A - Adverse Events not Monitored/Assessed
Description: Study not completed.
Arm/Group | 10% Phenylephrine
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03615508/Prot_SAP_000.pdf